CLINICAL TRIAL: NCT05396755
Title: Biliary Interventions in Critically Ill Patients With Secondary Sclerosing Cholangitis - a Multicenter, Randomized Controlled, Parallel Group Trial
Brief Title: Biliary Interventions in Critically Ill Patients With Secondary Sclerosing Cholangitis (BISCIT)
Acronym: BISCIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to insufficient recruitment.
Sponsor: Hannover Medical School (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BISCIT
Record Dates: First submitted 2022-05-03; First posted 2022-05-31 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Secondary Sclerosing Cholangitis
Keywords: biliary intervention; endoscopic therapy; endoscopic retrograde cholangiography

STUDY DESIGN:
Intervention Model Description: randomized, open-label, controlled, parallel group, multicenter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): The intervention group undergoes scheduled invasive evaluation of the biliary tract with endoscopic retrograde cholangiography (ERC) with biliary interventions (i.e. therapeutic ERC) every 8 weeks for 6 months.
  Interventions: Procedure: Endoscopic retrograde cholangiography (ERC)
- control (No Intervention): The control group receives non-interventional standard of care.

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiography (ERC) — invasive evaluation of the biliary tract with ERC and endoscopic interventions every 8 weeks until 6 months (24 weeks)
  Arms: interventional

SUMMARY:
This is a randomized, open-label, controlled, parallel group, multicenter clinical trial. Patients with confirmed secondary sclerosing cholangitis (SSC-CIP) will be randomized either in the intervention group undergoing scheduled invasive evaluation of the biliary tract or in the control group treated with non-interventional standard of care to demonstrate that programmed endoscopic therapy compared to a conservative strategy reduces the occurrence of treatment failures.

ELIGIBILITY:
Inclusion Criteria:

Patients have to fulfill all of the following inclusion criteria to be eligible for participation in this study:

1. Men, women*, inter/divers, age ≥18 and ≤ 80 years (conscious or unconscious patients may be included)
2. Signed written informed consent obtained by patient or legal representative in case of unconscious patient
3. Willingness to comply with treatment and follow-up procedures
4. Suspected SSC-CIP = episode of critical illness and intensive care unit treatment > 3 days within last 12 months
5. SSC-CIP is confirmed by ERC, (if the first ERC is performed at baseline, the patient may be considered as screening failure if the diagnosis is not confirmed)
6. Elevation of bilirubin ≥ 2.5 upper limit of normal (ULN) at Screening
7. Elevation of alkaline phosphatase (AP) or gamma-glutamyl-transferase (GGT) > 2.5 ULN or elevation of both at Screening
8. *Women without childbearing potential defined as follows:

   * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
   * hysterectomy or uterine agenesis or
   * ≥ 50 years and in postmenopausal state > 1 year or
   * < 50 years and in postmenopausal state > 1 year with serum Follicle Stimulating Hormone (FSH) > 40 IU/l and serum estrogen < 30 ng/l or a negative estrogen test, both at screening or

     *Women of childbearing potential:
   * who are practicing sexual abstinence (periodic abstinence and withdrawal are not acceptable) or
   * who have sexual relationships with female partners only and/or with sterile male partners or
   * who are sexually active with fertile male partner, have a negative pregnancy test during screening and agree to use reliable methods of contraception (failure rate of < 1% per year) from the time of screening until end of the clinical trial.

Exclusion Criteria:

1. Patient is too unstable to undergo ERC
2. Inclusion in any other intervention trial within the last 30 days
3. Pregnancy or lactation period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
occurrence of death | up to week 48
  The primary endpoint is the failure rate defined as a composite endpoint consisting of
  * occurrence of death or
  * necessity of liver transplantation or
  * occurrence of cholangiosepsis (defined by SEPSIS-3 criteria and diagnosis of acute cholangitis according to the Tokyo Guidelines), whatever occurs first.
necessity of liver transplantation | up to week 48
  The primary endpoint is the failure rate defined as a composite endpoint consisting of
  * occurrence of death or
  * necessity of liver transplantation or
  * occurrence of cholangiosepsis (defined by SEPSIS-3 criteria and diagnosis of acute cholangitis according to the Tokyo Guidelines), whatever occurs first.
occurrence of cholangiosepsis (defined by SEPSIS-3 criteria and diagnosis of acute cholangitis according to the Tokyo Guidelines), whatever occurs first. | up to week 48
  The primary endpoint is the failure rate defined as a composite endpoint consisting of
  * occurrence of death or
  * necessity of liver transplantation or
  * occurrence of cholangiosepsis (defined by SEPSIS-3 criteria and diagnosis of acute cholangitis according to the Tokyo Guidelines), whatever occurs first.

SECONDARY OUTCOMES:
Laboratory parameters (bilirubin in µmol/L) as change from baseline | week 24
Laboratory parameters (alkaline phosphatase in U/L) as change from baseline | week 24
Laboratory parameters (gamma-glutamyltransferase) as change from baseline | week 24
Laboratory parameters (aspartate aminotransferase in U/L) as change from baseline | week 24
Laboratory parameters (alanine aminotransferase in U/L) as change from baseline | week 24
Laboratory parameters (lactate dehydrogenase in U/L) as change from baseline | week 24
Laboratory parameters (glutamate dehydrogenase in U/L) as change from baseline | week 24
Laboratory parameters (creatinine in µmol/L) as change from baseline | week 24
Laboratory parameters (c-reactive protein in mg/L) as change from baseline | week 24
Laboratory parameters (cholinesterase in kU/L) as change from baseline | week 24
To analyze course of liver function (Model for endstage liver disease score as changes from baseline) | week 24
  Model for End-Stage Liver Disease (MELD) score 0-40 points with higher values indicating increasing impairment of liver function
Occurrence of unplanned Intensive care unit (ICU) admissions (necessity and days free of: intensive care unit care, invasive ventilation, renal replacement therapy, vasopressors within 6 months) | week 24
To analyze the need for anti-infective therapy (antibiotic treatment) in the different study arms | week 24
  Necessity of treatment with anti-infective medication (= treament with antibiotic oral or intravenously for acute cholangitis) (yes/no)
Occurrence of unplanned hospital admissions (necessity and days free of hospital care within 6 months) | week 24

OTHER OUTCOMES:
Changes in specific signatures in biliary microbiome | day1, week 8, week 16, week 24
To analyze the extent of biliary tract damage at magnetic resonance cholangiopancreatography (MRCP) in the different study arms. | week 24
  Extent of bile duct damage at 6-months MRCP compared to baseline as determined by central radiology reading
Occurrence of infections: cholangitis, cholecystitis | up to week 48
Occurrence of ERC-related complications: bleeding, perforation, pancreatitis, cholangitis, | day1, week 8, week 16, week 24
occurrence of serious adverse events | day1, week 8, week 16, week 24, week 32, week 40, week 48
  population

CONTACTS AND LOCATIONS:
Overall Officials: Hans H. Wedemeyer, Prof., Principal Investigator — Hannover Medical School, Department of Gastroenterology, Hepatology and Endocrinology
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stahl K, Klein F, Voigtlander T, Grosshennig A, Book T, Muller T, Wree A, Kuellmer A, Weigt J, Dechene A, Wedi E, Kandulski A, Lange CM, Holzwart D, von Witzendorff D, Ringe KI, Wedemeyer H, Heidrich B; BISCIT Study group. BISCIT: Biliary interventions in critically ill patients with secondary sclerosing cholangitis-a study protocol for a multicenter, randomized, controlled parallel group trial. Trials. 2023 Mar 31;24(1):247. doi: 10.1186/s13063-023-07260-w. PMID 37004078